CLINICAL TRIAL: NCT06556719
Title: Hoosier Sport Re-Social: A Biobehavioral Intervention in Rural Indiana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kyle A. Kercher, Assistant Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21473
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: CVD; Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hoosier Sport Re-Social Participants (Experimental): Arm will receive 6-weeks of intervention, including enhanced PE and health class curriculum
  Interventions: Behavioral: Hoosier Sport Re-Social
- Regular Health and PE Participants (No Intervention): Arm will receive regular PE and health class curriculum

INTERVENTIONS:
Behavioral: Hoosier Sport Re-Social — Hoosier Sport Re-Social is a 6-week school-based intervention designed to reduce cardiovascular disease risk in rural children. It includes twice-weekly physical activity sessions during PE classes and weekly social media literacy training in health classes, promoting healthier physical and digital behaviors.
  Arms: Hoosier Sport Re-Social Participants

SUMMARY:
Hoosier Sport Re-Social is a sport-based intervention designed to increase physical activity (PA) and reduce social media use among children in under-resourced rural areas, aiming to mitigate cardiovascular disease (CVD) risk. The intervention integrates physical activity with social media literacy (SML) training, addressing the dual challenges of low PA levels and high social media usage, which are prevalent in rural communities.

DETAILED DESCRIPTION:
Hoosier Sport Re-Social is a comprehensive, sport-based intervention designed to address the dual challenges of low physical activity (PA) and high social media use among children in under-resourced rural areas. This innovative program aims to reduce cardiovascular disease (CVD) risk by promoting healthier behaviors through the integration of physical activity and social media literacy (SML) training. Recognizing that CVD is a leading cause of death, particularly in under-resourced populations, and that fewer than one in five U.S. children meet the recommended PA levels-especially in rural areas-this intervention targets a significant public health need.

The program is designed to be implemented within the school setting, leveraging both physical education (PE) and health classes to deliver its core components. The PA portion of the intervention takes place during PE classes, where students engage in structured sport activities aimed at increasing daily physical activity levels. This component is designed to enhance students' fitness, build confidence in their physical abilities, and foster a lifelong interest in staying active.

Complementing the physical activity focus, the SML portion is integrated into health classes. Here, students are educated about the impacts of social media on health, particularly its role in influencing behavior and well-being. The curriculum equips students with the knowledge and skills to critically analyze social media content, make informed decisions about their digital consumption, and develop healthier online habits.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in 7th-9th grade
* provides parental consent
* provides assent

Exclusion Criteria:

- Inability to attend school regularly during the 6-week intervention period

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | Measured at week 0 and week 6
  How feasible the intervention was from the perspective of the participants. This is measured through questionnaire.
Acceptability of Intervention Measure (IAM) | Measured at week 0 and week 6
  How acceptable the intervention is to the participants. This is measured through questionnaire.
Intervention Appropriateness Measure (AIM) | Measured at week 0 and week 6
  How appropriate the intervention is to the participants. This is measured through questionnaire.

SECONDARY OUTCOMES:
Daily Total Physical Activity of Participants | Week 1 (for 7 days), and week 6 (for 7 days)
  Accelerometers (Axivity - AX3 model) will be used to track total daily physical activity
Heart Rate of Participants | HR will be taken at week 0 and week 6 before and following the 6-minute walk test.
  heart rate measured via a blood pressure monitor
Blood Pressure of Participants | BP will be taken at week 0 and week 6 before and following the 6-minute walk test.
  Blood pressure measured via a blood pressure monitor
Basic Psychological Needs of Participants in Intervention Environment | Assessed at week 0 and week 6
  Basic Psychological Needs and Satisfaction and Frustration scale. This entails feelings/perceptions of autonomy, relatedness, competence, enjoyment, satisfaction, and frustration in the study setting. Higher scores indicate greater satisfaction.
Physical Literacy of Participants | Assessed at week 0 and week 6
  the Canadian Assessment of Physical Literacy second addition (CAPL-2) will be used. A higher score on the CAPL-2 indicates higher physical literacy.
Cardiovascular Fitness Levels of Participants | Assessed at week 0 and week 6
  the 6-minute walk test will be used to assess changes in fitness. Greater distance walked in the 6 minute time frame is related to greater levels of cardiovascular fitness.
Muscular Endurance Levels of Participants | Assessed at week 0 and week 6
  The plank test will be used to assess changes in fitness. The longer the plank is held, the greater the muscular endurance of the participant.
Daily screen time | Assessed at week 0 and week 6
  data from participants' phone settings will be used to capture daily screen time. Participants will navigate to their screen time settings, where a comprehensive and objective report of their weekly screen time (including average daily screen time) is available. Here, participants will screenshot this data and airdrop it to a secured IU dropbox location.
Daily social media usage | Assessed at week 0 and week 6
  data from participants' phone settings will be used to capture daily screen time. Participants will navigate to their screen time settings, where a comprehensive and objective report of their weekly screen time (including average daily social media usage) is available. Here, participants will screenshot this data and airdrop it to a secured IU dropbox location.
Social media addiction | Assessed at week 0 and week 6
  participants will complete the Bergen Social Media Addiction Scale to assess social media addiction.
Inhibitory control | Assessed at week 0 and week 6
  The Color-Word trial from the Stroop Color and Word Test will be delivered on an iPad/tablet to participants to measure inhibitory control.
Body Satisfaction | Assessed at week 0 and week 6
  The Body Satisfaction Questionnaire (BSQ) will be completed to assess participants satisfaction of their body shape.
Body Appreciation | Assessed at week 0 and week 6
  The Body Appreciation Scale (version 2) (BAS-2) will be completed to assess participants' appreciation of their bodies.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Kercher, PhD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University, Bloomington, Indiana
  - White River Valley Middle School, Lyons, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watkins JM, Goss JM, Kercher VMM, Coble CJ, Werner NE, Weaver RG, Kercher KA. Hoosier Sport Re-Social: a protocol for developing a biopsychosocial body satisfaction intervention in rural Indiana. Pilot Feasibility Stud. 2025 Aug 25;11(1):113. doi: 10.1186/s40814-025-01695-5. PMID 40855334